CLINICAL TRIAL: NCT01754415
Title: Evaluation of Exercise Benefits to Promote Health Aging Among Chronically Ill Geriatrics in a Community.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: FEMH-IRB-098101-3
Record Dates: First submitted 2012-11-06; First posted 2012-12-21 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes; Hypertension; Osteoporosis; Osteoarthritis
Keywords: Aging; Chronic illness; Resistance circuit training
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Osteoporosis; Osteoarthritis; Chronic Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (No Intervention): Do exercise at home with video program designed by our team.
- hydraulic resistance circuit training (Experimental): Intervention:12 weeks resistance training
  Interventions: Device: hydraulic resistance circuit training

INTERVENTIONS:
Device: hydraulic resistance circuit training — 12 weeks (3 times per week, 40 min circuit) of hydraulic resistance circuit training that consisted of 10 types of equipments for different part of strength training.
  Arms: hydraulic resistance circuit training

SUMMARY:
The aim of this study is to evaluate the effect of hydraulic resistance circuit training for elderly people with chronic illness.

DETAILED DESCRIPTION:
This study is divided into three years. The aim of the first year is to analyze the types and percentage of chronic illness in middle- and old-aged population in communities and the impact on their physical and mental function. The Second year, we will use proper exercise prescriptions with exercise equipment available for chronic illness population and examine the improvement of their physical and mental functions after exercise intervention. The third year, we will adopt the concept of social marketing to promote knowledge about health-related fitness and exercise to communities and help to establish exercise center. To chronic illness people, the study seeks to delay the progression of disease and disability by encouraging them to participate in prescribed exercises. To relatively healthy people, exercise can achieve the purposes of healthy aging, decreased chronic illness, and improved ADLs function and life quality.

ELIGIBILITY:
Inclusion Criteria:

Subjects were recruited at the age of 45-80, and can communicate verbally and in writing.

Exclusion Criteria:

Subjects had physical limitation in sports and were advised not to exercise by doctors.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) | three years
  Level of self-reported physical activity assessed with the International Physical Activity Questionnaire,IPAQ and expressed as MET-minutes.

SECONDARY OUTCOMES:
Body composition measurement | three years
  Body composition refers to the amount of relative fat to muscle you have in your body, which the items include height (cm), weight(kg), body mass index (BMI), muscle mass(kg), fat (%), fat mass, fat free mass (FFM), and total body water (TBW).
The physical fitness assessment | three years
  The physical fitness designed to evaluate several components of functional ﬁtness was as follows:
  30-second chair stand test: Count the times that person rises in 30-s without pushing off with the arms.
  Chair sit and reach: Measure the distance with an 20-cm ruler that a person is short of reaching the toe (minus score) or beyond the toe (plus score).
  2-minute step test: Determine the times that person can step in place, raising (Alternate test) the knees to a height halfway between the iliac crest and middle of the patella, in 2-min.
  Back scratch: Measure the distance between (or the overlap of) the middle ﬁngers behind the back when trying to touch the middle ﬁngers of both hands together behind the back.
  8-foot up and go: Measure the time it takes to get out of a chair, walk 8-feet to and around a cone, and return to the chair.

CONTACTS AND LOCATIONS:
Overall Officials: Tsung-Ching Lin, Master, Study Chair — Far Eastern Memorial Hospital
Locations (1):
- Tsung-Ching Lin, New Taipei City, Taiwan, Taiwan